CLINICAL TRIAL: NCT01924273
Title: Novel Treatment for Port Wine Stain Birthmarks
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Kristen Kelly M.D.,Professor Departments of Dermatology and Surgery, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20139337
Record Dates: First submitted 2013-07-17; First posted 2013-08-16 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Port-Wine Stain
Keywords: Port Wine Stain Birthmarks
MeSH Terms: conditions — Port-Wine Stain | interventions — Talaporfin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Port Wine Stain Birthmarks (Other): Combined Photodynamic/Pulsed Dye Laser Therapy/Talaporfin sodium
  Interventions: Drug: Talaporfin sodium

INTERVENTIONS:
Drug: Talaporfin sodium — Combined Photodynamic/Pulsed Dye Laser Therapy/Talaporfin sodium
  Other Names: Combined Laser treatment andTalaporfin sodium

SUMMARY:
Port wine stains Birthmark are congenital, progressive vascular malformations of the skin that occur in approximately 0.7% of newborns. Approximately 1.5 million individuals in the United States and 32 million people worldwide have Port wine stains birthmarks. Two-thirds of these malformations occur on the face. Personality development of virtually all patients is adversely affected as a result of the negative reaction of others to a "marked" person. Detailed studies have documented lower self-esteem and difficulties with interpersonal interactions in Port wine stains patients. Port wine stains are initially flat and red, but with time, they tend to darken to purple and become thickened as vascular nodules develop. This thickening occurs in approximately two-thirds of lesions and further disfigures the facial features of many patients.

DETAILED DESCRIPTION:
Pulsed dye laser is currently the standard of care treatment for Port wine stains. Researchers at University of California Irvine at Beckman Laser Institute Medical Clinic can use Photodynamic therapy, another treatment option for Port wine stains. Photodynamic therapy involves light activation of a photosensitizer (a drug that is responsive to light or radiant energy). Because the photosensitizer can be localized to a desired portion of the Port wine stain, Photodynamic therapy creates an opportunity for targeted destruction of Port wine stains.

Researchers will use a photosensitizer medication called Talaporfin sodium, an intravenously administered investigational photosensitizer, being evaluated for multiple clinical indications. Photodynamic therapy with talaporfin sodium has been investigated for many different conditions, and can be used for treatment for Port wine stains. Photosensitivity precaution instructions will be provided, including appropriate photo protective clothing, protective hat and sunglasses that wrap around the temples to help minimize lateral sun light exposure when traveling home following discharge from the study site.

For efficacy, evaluated study variable will be Port wine stain blanching, and the researchers can use diffuse reflectance imaging chromametry, Laser Speckle Imaging and Spatial Frequency Domain Imaging to measure the change of Port wine stain blanching. The maximum power of the Laser Speckle Imaging and Spatial Frequency Domain Imaging light source is 10-50 mW, which is comparable to halogen-bulb household flashlights. Efficacy will be evaluated based on comparison of pre-treatment visit and post treatment day 1, week 1, week 4, and week 12 measurements.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female 18 years and older
* Have Port Wine Stain Birthmarks non-facial

Exclusion Criteria:

* Under 18 years of age
* No Port Wine Stain Birthmarks
* pregnant/breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-06; Primary Completion 2017-07-03 (Actual); Study Completion 2017-07-03 (Actual)

PRIMARY OUTCOMES:
Port wine stain blanching | up to 12 weeks
  The outcome measure will be PWS blanching as assessed by Diffuse Reflectance Imaging/Laser Speckle Imaging/Spatial Frequency Domain Imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Kelly, MD, Principal Investigator — Beckman Laser Institute
Locations (1):
- Beckman Laser Institute, Irvine, California, United States